CLINICAL TRIAL: NCT01457547
Title: Study to Assess and Compare the Immunogenicity and Reactogenicity of GlaxoSmithKline Biologicals' DTPa-HBV-IPV/Hib Vaccine (INFANRIX™ HEXA) and Aventis Pasteur MSD's DTPa-HBV-IPV-Hib Vaccine (HEXAVAC™) Given at 3, 5 and 11-12 Months of Age
Brief Title: Comparison of Immunogenicity and Reactogenicity of INFANRIX™ HEXA and HEXAVAC™ Vaccines as a Primary Vaccination Course
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 217744/094
Record Dates: First submitted 2011-10-13; First posted 2011-10-24 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis B; Poliomyelitis; Diphtheria; Acellular Pertussis; Tetanus; Haemophilus Influenzae Type b
Keywords: HEXAVACTM; InfanrixTM HEXA; DTPa-HBV-IPV-Hib; DTPa-HBV-IPV/Hib
MeSH Terms: conditions — Hepatitis B; Poliomyelitis; Diphtheria; Tetanus; Haemophilus Infections | interventions — Hexavac

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- DTPa 1 Group (Experimental)
  Interventions: Biological: DTPa-HBV-IPV/Hib Vaccine (INFANRIX™ HEXA)
- DTPa 2 Group (Active Comparator)
  Interventions: Biological: DTPa-HBV-IPV-Hib vaccine (HEXAVAC™)

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib Vaccine (INFANRIX™ HEXA) — Three doses administered intramuscularly
  Arms: DTPa 1 Group
Biological: DTPa-HBV-IPV-Hib vaccine (HEXAVAC™) — Three doses administered intramuscularly
  Arms: DTPa 2 Group

SUMMARY:
The study will compare the immunogenicity and the reactogenicity of INFANRIX™ HEXA and HEXAVAC™ vaccines in a 3, 5 and 11 - 12 month vaccination schedule.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female subject between 8 and 15 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject prior to the study entry.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a normal gestation period between 36 and 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B and/or Hib vaccination or disease.
* Planned administration of a vaccine not foreseen by the study protocol since birth and during the period starting 30 days before the administration of the first dose and ending 30 days after the last dose of the three-dose primary vaccination course, with the exception of licensed Neisseria meningitides conjugate vaccines or Bacillus Calmette-Guérin (BCG) vaccine that can be given in between study visits or after the third visit, provided they are given preferably with a 4 weeks interval but not less than 3 weeks apart from the study vaccine doses.
* Chronic administration or planned administration of immuno-suppressants or other immune-modifying drugs since birth.
* Planned administration of immunoglobulins and/or any blood products since birth or planned administration during the period up to 30 days after the third dose of the primary vaccination course.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of seizures, progressive neurological disease or intra-cerebral haemorrhage.
* Major congenital defects or serious chronic illness.
* Acute febrile illness at the time of planned vaccination
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.

Ages: 8 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 494 (Actual)
Dates: Start 2003-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccine in terms of antibody concentrations | Prior to the third primary vaccination dose ( Months 8-9)

SECONDARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccine in terms of antibody concentrations | One month after the second and third primary vaccination dose (Month 3 and Months 9-10)
Immunogenicity with respect to the components of the study vaccine in terms of number of seroprotected subjects defined by antibody concentration | Prior to and one month after the third primary vaccination dose ( Months 8-9 and Months 9-10)
Immunogenicity with respect to the components of the study vaccine in terms of number of seropositive subjects | Prior to and one month after the third primary vaccination dose ( Months 8-9 and Months 9-10)
Occurrence of solicited symptoms | Within 4 days (Day 0 -Day 3) after each vaccine dose
Occurrence of a grade "3" solicited symptoms | Within 4 days (Day 0 -Day 3) after each vaccine dose
Occurrence of unsolicited adverse events | Within 31 days after any vaccination
Occurrence of Serious Adverse Events | Throughout the entire study up to (Month 0 to Month 9-10) and including 30 days after last vaccination (Month 9-10)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Helsinki, Finland
- Italy (6):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Galatina (LE), Apulia
  - GSK Investigational Site, Maglie (LE), Apulia
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Sassari, Sardinia
- Sweden (2):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Örebro

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kilpi et al. Comparison of the immunogenicity and reactogenicity of two hexavalent DTPa-HBV-IPV/Haemophilus influenzae type b vaccines administered at 3, 5 and 11-12 months of age. Abstract presented at the 24th annual meeting of the European Society for Paediatric Infectious Diseases (ESPID), Basel Switzerland 03-05 May, 2006.
- [Background] Kilpi TM, Silfverdal SA, Nilsson L, Syrjanen R, Belloni C, Desole M, Triban C, Storsaeter J, Soila M, Jacquet JM. Immunogenicity and reactogenicity of two diphtheria-tetanus-acellular pertussis-hepatitis B-inactivated polio virus-Haemophilus influenzae type b vaccines administered at 3, 5 and 11-12 months of age. Hum Vaccin. 2009 Jan-Feb;5(1):18-25. doi: 10.4161/hv.5.1.6369. Epub 2009 Jan 2. PMID 18690013
- [Background] Van Der Meeren O, Kuriyakose S, Kolhe D, Hardt K. Immunogenicity of Infanrix hexa administered at 3, 5 and 11 months of age. Vaccine. 2012 Apr 5;30(17):2710-4. doi: 10.1016/j.vaccine.2012.02.024. Epub 2012 Feb 18. PMID 22349525
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 217744/094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register